CLINICAL TRIAL: NCT02782988
Title: Assesment of Olfactory Disorders and Performance of a New Olfactory Test in Children With Congenital Cytomegalovirus Infection
Brief Title: Assesment of Olfactory Disorders and Performance of a New Olfactory Test in Children With Congenital CMV
Acronym: INFECSMELL
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-091
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Olfaction; CMV
MeSH Terms: conditions — Cytomegalovirus Infections; Anosmia | interventions — Otoacoustic Emissions, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CMV symptomatic at birth: olfactory tests, otoacoustic emissions (OAE)
  Interventions: Other: olfactory tests, otoacoustic emissions (OAE)
- CMV asymptomatic at birth: olfactory tests, otoacoustic emissions (OAE)
  Interventions: Other: olfactory tests, otoacoustic emissions (OAE)
- Healthy controls: olfactory tests, otoacoustic emissions (OAE)
  Interventions: Other: olfactory tests, otoacoustic emissions (OAE)

INTERVENTIONS:
Other: olfactory tests, otoacoustic emissions (OAE) — Two series of olfactory tests will be performed : 1) the first one with simple odorants and 2) the second one with binary mixtures of odorants. These tests of nasal chemosensory performance are based on pen-like odor dispensing devices (Sniffin' Sticks, Burghardt, Wedel, Germany) and measure odor discrimination ability of young children in less than 15 min.

SUMMARY:
CMV lesions were found in the olfactory system of children with congenital CMV infection but no study has hitherto examined the impact of congenital CMV infection on olfaction. So the investigators propose in this study to assess the proportion of children with olfactory deficits among children with congenital CMV infection. Second this study will also evaluate performances of a new olfactory test, based on discrimination of binary odorant mixtures.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the first cause of congenital deafness resulting from viral infection. Hearing loss may occur several years after birth in childhood and be often progressive. Detection of hearing impairment is of major interest for children because it will allow the early use of a hearing aid minimizing the impact of these deficits on the cognitive development.

The study hypothesis is that a link might exist between hearing deficits and olfactory deficits in these children due to viral lesions on the two sensory systems. Thus early exploration of olfaction might allow early detection of starting deterioration of hearing or predict the occurrence of deafness. Moreover, this exploration is easy, non invasive, fast to set up and adapted to very young children. No study has hitherto assessed the impact of congenital CMV infection on olfaction.

The proportion of children with olfactory deficits will be assessed among children with congenital CMV infection, using parts of a discrimination test of simple odorants (Sniffin' Sticks, Burghardt, Wedel, Germany). The performances of a new olfactory test developed by the investigators that uses binary mixtures of odorants, will also be assessed. These tests of nasal chemosensory performance are based on pen-like odor dispensing devices and measure odor discrimination ability of young children in less than 15 min. Finally, this study aims at demonstrate, if it exists, the association between olfactory deficits and hearing loss in children with congenital CMV infection.

This study will be conducted in 80 patients and 40 healthy subjects (3-10years). The healthy children will be matched for age and gender. Selection will be made based on medical records during the course of standard care visit. After collection of informed consent, olfactory tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 3 years old and ≤ 10 years old
* Oral consent of the child to participate in the study
* Written informed consent of the two parents
* Congenital CMV infection : 1) asymptomatic form at birth and 2) symptomatic form at birth. The latter is defined by the presence of at least one of the following clinical signs: growth retardation, prematurity,petechiae, splenomegaly, thrombocytopenia, jaundice, low number of platelets, ictere, digestive disorders ...

NOTE: CMV diagnosis is made on the following criteria: positive CMV PCR in urine and / or blood in the first 3 weeks of life or retrospective diagnosis on the presence of a positive PCR on the Guthrie test performed at 3-7 days of life.

Exclusion Criteria:

* Medical care incompatible with the objective of the study,
* Patient who would object to the protocol
* No clinical condition that may interfere with the study, e.g.: no chronic sinusitis, nasopharyngitis, etc.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 80 children with congenital CMV infection will be included in a monocentre study : 40 children which symptomatic CMV infection at birth and 40 children with asymptomatic form of infection at birth. To evaluate the performance of the new olfactory test, 40 controlled healthy children matched for age and gender will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Percentage of children with olfactory disorders among children with congenital CMV infection. | Inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Françoise LAZARINI, PhD, Study Director — Institut Pasteur, Paris France
Locations (2):
- France (2):
  - Hopital Bicêtre, Le Kremlin-Bicêtre
  - Robert Debré Hospital, Paris

IPD SHARING:
Plan to Share IPD: No